CLINICAL TRIAL: NCT06219421
Title: Automatic Phenotyping of Patients on 2D Photography
Acronym: AIDY2
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AIDY 2
Record Dates: First submitted 2023-12-28; First posted 2024-01-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Dysmorphia; Orphan Diseases; Dysmorphies Craniofaciales
Keywords: artificial intelligence
MeSH Terms: conditions — Congenital Abnormalities; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Clinical data reuse
- Controls
  Interventions: Other: Clinical data reuse

INTERVENTIONS:
Other: Clinical data reuse — Clinical data reuse

SUMMARY:
The field of artificial intelligence is booming in medicine and in the field of diagnosis. The data can be varied: x-rays, pathology sections, or photographs.

It is considered that 30 to 40% of the 7000 rare diseases described to date cause craniofacial dysmorphia. Their detection sometimes requires the trained eye of a geneticist, because certain phenotypic traits are subtle. These diagnostic difficulties and the fact that certain diseases are extremely uncommon lead to considerable diagnostic delays

ELIGIBILITY:
The patient inclusion criteria are:

* Patients followed in medical genetics,
* Patients undergoing maxillofacial surgery, or craniofacial surgery as part of the management of a pathology, of genetic origin or not, associated with dysmorphism of the head and neck,
* Patients for whom frontal and profile facial photographs are taken as part of their treatment.

The inclusion criteria for control subjects are:

* Patients followed in maxillofacial surgery, for a disease other than a rare disease associated with dysmorphia in the head or neck: acute pathology (wound) or chronic (gynecomastia).
* Patients for whom frontal and profile facial photographs are taken as part of their treatment.

The criteria for non-inclusion of patients are:

* Patients who have undergone facial or skull surgery before the first photo was taken.
* Person subject to a judicial safeguard measure.
* People objecting to the reuse of their health data.

The criteria for non-inclusion of control subjects are:

* Pathologies affecting facial symmetry (dental cellulitis, displaced fractures).
* Patient followed for dysmorphic syndrome or in whom dysmorphic syndrome has been suspected.
* Person subject to a judicial safeguard measure.
* People objecting to the reuse of their health data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment will be carried out either:
  In Necker in the services of:
  * Medical genetics
  * Maxillofacial surgery / plastic surgery
  * Neurosurgery (functional craniofacial surgery unit)
  Outside Necker:
  * In other national university hospitals: Lille (maxillofacial surgery department), Nantes (maxillofacial surgery department), Montpellier (clinical genetics department)
  * In other international university hospitals: London (GOSH, London, Professor Dunaway) and Bangkok (genetics department, Professor Porntaveetus)
  * In a private orthodontic practice
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Learning an algorithm on 2D front and profile photographs, by extracting geometric and textural features, to help the practitioner carry out a diagnosis. | through study completion, an average of 1 year
  Learning an algorithm on 2D front and profile photographs, by extracting geometric and textural features, to help the practitioner carry out a diagnosis.

SECONDARY OUTCOMES:
Carry out phenotype/genotype correlations to explain the phenotype of a particular genetic variant | through study completion, an average of 1 year
  Carry out phenotype/genotype correlations to explain the phenotype of a particular genetic variant
Study the facial characteristics of a syndrome depending on ethnicity | through study completion, an average of 1 year
  Study the facial characteristics of a syndrome depending on ethnicity
Study the facial characteristics of a syndrome depending on age | through study completion, an average of 1 year
  Study the facial characteristics of a syndrome depending on age

CONTACTS AND LOCATIONS:
Locations (1):
- Necker - Hôpital des Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No